CLINICAL TRIAL: NCT05208723
Title: Stress and Emotion Management Training for Female Entrepreneurs in Ethiopia
Brief Title: Addressing Stress Amongst Female Entrepreneurs in Addis Ababa, Ethiopia: a Pilot Study
Acronym: DWMTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: World Bank (Other)
Collaborators: Ethiopian Medical Association (Unknown); Addis Ababa University (Other); PSI Ethiopia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DWMTS
Record Dates: First submitted 2021-12-20; First posted 2022-01-26 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Stress, Psychological; Emotion Regulation; Social Psychology; Economic Problems; Mental Stress
Keywords: Stress management; Economic benefits; Mental health
MeSH Terms: conditions — Stress, Psychological; Emotional Regulation; Psychological Well-Being | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Enrolled participants are randomized to intervention or control group
Who Masked: Investigator
Masking Description: Randomized using computer generated randomization at one point in time by an independent researcher
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress and emotion management (Experimental): A locally adapted self-help guidebook originally developed by the World Health Organization (WHO), 'Doing what matters in times of stress' for managing disruptive emotions and psychological distress, will be delivered to female entrepreneurs at their residence, followed by 5-6 phone calls from a trained mental health helper to reinforce the materials over a 6-week period. The intervention is intended to help people manage their psychological distress associated with a range of adversities but is not intended for participants with severe mental health problems such as psychosis or imminent risk of suicide.
  Interventions: Behavioral: Stress and emotion management
- Control group (No Intervention): No intervention. May receive intervention post study if findings are indicative of any benefit.

INTERVENTIONS:
Behavioral: Stress and emotion management — The handbook materials and lay helper scripts are based on principles of Acceptance and Commitment Therapy (ACT), and aims to enhance psychological flexibility. Psychological flexibility reflects how a person adapts to fluctuating situational demands, reconfigures mental resources, shifts perspective, and balances competing needs. ACT teaches alternative methods to accommodate difficult thoughts and feelings, primarily through mindfulness techniques. At the same time, ACT also focuses on guiding participants to live in ways consistent with their personal values.
  Other Names: Doing what matters in times of Stress; Acceptance and Commitment Therapy (ACT)
  Arms: Stress and emotion management

SUMMARY:
The overall objective of this study is to evaluate the impact of the "Doing What Matters in Times of Stress Guided Self-Help" handbook along with lay helper session on managing stress and emotion on mental distress and well-being. If successful, the study will assess its impact on business performance among women entrepreneurs in Ethiopia.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the impact of the "Doing What Matters in Times of Stress Guided Self-Help Manual" on mental distress and if successful, see its impact on business performance among women entrepreneurs in Ethiopia. The study will be conducted in Addis Ababa, Ethiopia. A pilot randomized controlled trial (RCT) will be conducted to investigate the impact of the "Doing What Matters in Times of Stress Guided Self-Help Manual" intervention to reduce psychological distress and functional impairment among women entrepreneurs in Ethiopia. The investigators will screen approximately1200 women over the phone and identify 200 eligible women for the study. An in-person baseline survey will be conducted with the 200 eligible women and the participants will be randomized (using computer generated randomization) to either the doing what matters in times of stress self-help manual intervention (n=100) or wait list control (n=100). This will be followed by 6 phone-based sessions over 6-8 weeks to review handbook materials for the intervention group only. After six weeks, phone-based follow-up survey will be conducted with participants in both the intervention and control groups. If the intervention is found to be effective in reducing distress or stress at follow-up assessment, then the baseline survey will be repeated at 6-9 months post intervention both for the intervention and control group participants. Additionally, based on findings from the pilot study a larger sample of participants will be screened and enrolled (approximately 1000 women) and randomized to the intervention or wait-list control arm to be followed up at 6-9 months post intervention. The primary outcomes for this study will be psychological distress. Participants' performance on their businesses and self-esteem will be secondary outcomes for the study. A generalized linear model with appropriate statistical specifications and accounting for baseline values and any imbalanced variables at baseline (where available) will be used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18;
* Women entrepreneurs who obtained loan or business skills training from WEDP;
* Those who have plan to live in Addis Ababa in the next six months;
* Those who can read and speak Amharic and can understand the study questionnaire;
* Those who have capacity to provide informed consent;
* Score 8 or above on the Ethiopian adaptation of Kessler-6;

Exclusion Criteria:

* Kessler 6 score >20;
* Those who have recent or current suicidal thoughts or plans;
* Those who have limitation to understand the study questionnaire;
* Those who have not capacity to provide informed consent;
* Do not own a mobile phone;
* Not interested in receiving the intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — identifying as women
Enrollment: 200 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mental Distress using the Kessler Psychological Distress Scale (K-6) | 4-6 weeks post intervention
  Minimum value of 0 and a maximum value of 24. Higher scores indicate high levels of psychological distress (worse outcome)
Mental Distress using the Kessler Psychological Distress Scale (K-6) | 6-9 months post intervention
  Minimum value of 0 and a maximum score of 24. Higher scores indicate high levels of psychological distress (worse outcome)
Depression using the Patient Health Questionnaire (PHQ-9) | 4-6 weeks post intervention
  Minimum score 0 and a maximum score of 27. Higher scores indicate increased levels of depressive symptoms (worse outcome).
Depression using the Patient Health Questionnaire (PHQ-9) | 6-9 months post intervention
  Minimum score 0 and a maximum score of 27. Higher scores indicate increased levels of depressive symptoms (worse outcome).
Stress using the Perceived Stress Scale | 4-6 weeks post intervention
  Minimum score of 0 and a maximum of 40. Higher scores indicate high levels of perceived stress (worse outcome). Investigators will reverse code items 4,5, 7 and 8
Stress using the Perceived Stress Scale | 6-9 months post intervention
  Minimum score of 0 and a maximum of 40. Higher scores indicate high levels of perceived stress (worse outcome). Investigators will reverse code items 4,5, 7 and 8
Self-reported Business outcomes | 6-9 months post intervention
  Self-reported past month profits in local currency

SECONDARY OUTCOMES:
Self-reported Business outcomes | 4-6 weeks post intervention
  Self-reported past month profits in local currency
Self-reported Business Closure | 4-6 weeks post intervention
  Self-reported business closure
Self-reported Business Closure | 6-9 months post intervention
  Self-reported business closure
Self-reported number of recent hires | 4-6 weeks post intervention
  Average self-reported number of employees hired in the past month
Self-reported number of employees | 6-9 months post intervention
  Average self-reported number of employees
Self-Esteem using the Rosenberg Self-esteem Scale | 4-6 weeks post intervention
  Minimum score 10 and a maximum score of 40. Investigators will reverse code items 3,5,8,9 and 10 . Higher scores indicate high levels of self-esteem (better outcome)
Self-Esteem using the Rosenberg Self-esteem Scale | 6-9 months post intervention
  Minimum score 10 and a maximum score of 40. Investigators will reverse code items 3,5,8,9 and 10. Higher scores indicate high levels of self-esteem (better outcome)
World Health Organisation- Five Well-Being Index (WHO-5) | 4-6 weeks post intervention
  Minimum score of 0 and a maximum of 25. Higher scores mean better wellbeing (better outcome). Scores are transformed to 0-100 (by multiplying by 4.
World Health Organisation- Five Well-Being Index (WHO-5) | 6-9 months post intervention
  Minimum score of 0 and a maximum of 25. Higher scores mean better wellbeing (better outcome). Scores are transformed to 0-100 (by multiplying by 4.
Functional Impairment using the World Health Organization Disability Assessment Schedule (WHODAS-2.0 -12 item version) | 6-9 months post intervention
  Minimum score of 12 and a maximum of 60. Higher scores indicate high levels of disability (worse outcome)
Functional Impairment using the World Health Organization Disability Assessment Schedule (WHODAS-2.0 -12 item version) | 4-6 weeks post intervention
  Minimum score of 12 and a maximum of 60. Higher scores indicate high levels of disability (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Naira Kalra, PhD, Principal Investigator — World Bank; Adiam Hailemicheal, MSc, Principal Investigator — World Bank; Kassahun Habtamu Mekonnen, PhD, Principal Investigator — Addis Ababa University; Medhin Selamu Tegegn, PhD, Principal Investigator — College of health science, Addis Ababa University, Ethiopia
Locations (1):
- PSI and World Bank, Ethiopia, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
All unidentified IPD that underlie results in a publication will be shared if doing so is approved by the Institutional Review Board and clears privacy and security requirements set by the World Bank microdata portal.
Time Frame: Post study in 2023. Will be shared for at least 2 years.
Access Criteria: Publicly available. Use of the dataset must be acknowledged using a citation which would include:
  * the Identification of the Primary Investigator
  * the title of the survey (including country, acronym and year of implementation)
  * the survey reference number
  * the source and date of download
URL: https://www.worldbank.org/en/programs/africa-gender-innovation-lab/brief/africa-gender-innovation-lab-data